CLINICAL TRIAL: NCT03894904
Title: Double-Blind, Randomized, Controlled Trial, Small Volume Bolus of Papaverine Versus Heparin to Maintain Patency of Peripheral Arterial Catheters in Pediatric Patients Undergoing Surgical Procedures: Pilot Study
Brief Title: Papaverine vs Heparin for Peripheral Arterial Catheter Patency in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nischal Krishamurthy Gautam, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC-MS-19-0059
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pediatrics; Anesthesia; Vasospasm
Keywords: Heparin; Papaverine
MeSH Terms: interventions — Papaverine; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Papaverine plus heparin during procedure, with rescue papaverine as needed (Experimental): 1 mL bolus of papaverine (0.12 mg/mL) plus heparin (2 units/mL) in saline (NaCl 0.9%) will be administered as soon as the arterial catheter is placed and secured, and a 1 mL bolus of papaverine (0.12 mg/mL) plus heparin (2 units/mL) in saline (NaCl 0.9%) will be administered one hour after initial bolus. If the arterial catheter spasm/patency or waveform does not improve 10 minutes after the second bolus, then the anesthesiology care team will consider treating clinically with 0.3 mg of papaverine.
  Interventions: Drug: Papaverine; Drug: Heparin; Drug: Rescue papaverine, as needed
- Heparin during procedure, with rescue papaverine as needed (Active Comparator): 1 mL bolus of heparin (2 units/mL) in saline (NaCl 0.9%) will be administered as soon as the arterial catheter is placed and secured, and a 1 mL bolus of heparin (2 units/mL) in saline (NaCl 0.9%) will be administered one hour after initial bolus. If the arterial catheter spasm/patency or waveform does not improve 10 minutes after the second bolus, then the anesthesiology care team will consider treating clinically with 0.3 mg of papaverine.
  Interventions: Drug: Heparin; Drug: Rescue papaverine, as needed

INTERVENTIONS:
Drug: Papaverine — 0.12 mg/mL papaverine administered as soon as the arterial catheter is placed and secured, and 0.12 mg/mL papaverine administered one hour after initial dose
  Arms: Papaverine plus heparin during procedure, with rescue papaverine as needed
Drug: Heparin — 2 units/mL heparin administered as soon as the arterial catheter is placed and secured, and 2 units/mL heparin administered one hour after initial dose
Drug: Rescue papaverine, as needed — If the arterial catheter spasm/patency or waveform does not improve 10 minutes after the second papaverine plus heparin or heparin only dose, then the anesthesiology care team will consider treating clinically with 0.3 mg of papaverine.

SUMMARY:
The purpose of this study is to compare intraoperative papaverine plus heparin to heparin alone for prevention of arterial spasm and maintenance of patency of peripheral arterial catheters during surgery in pediatric patients. The hypothesis is that periodic, intraoperative small-volume boluses of diluted papaverine plus heparin in peripheral arterial catheters of pediatric patients will prevent arterial spasm and help maintain patency of arterial catheters during general anesthesia.

DETAILED DESCRIPTION:
Peripheral arterial catheters measure blood pressure with every heartbeat and provide valuable information regarding the status of the heart and the overall well being. It is of utmost importance to maintain the utility and patency of these catheters throughout the procedure. As standard procedure, heparin, a blood thinner, is used routinely during the surgical procedure to keep these catheters from clotting, and papaverine, an arterial relaxation agent, is used after surgery to maintain patency of these catheters.

In this study, participants will be randomized to receive two boluses of papaverine with heparin during the procedure (experimental arm) or heparin alone during the procedure (control arm) [in both arms, the first bolus will be administered as soon as the arterial catheter is placed and secured and again one hour after initial bolus]. If the arterial catheter spasm/patency or waveform does not improve 10 minutes after the second bolus, then the anesthesiology care team will consider treating clinically with 0.3 mg of papaverine.

ELIGIBILITY:
Inclusion Criteria:

- All patients age 0-17 years who would require elective placements of arterial catheters based on patients clinical complexity (ex. congenital heart disease) or based on the type of surgery (ex. open heart surgery).

Exclusion Criteria:

* Patients with a history of significant liver dysfunction.
* Patients undergoing liver transplants.
* Patients with Grade 2 or more of intraventricular hemorrhage.
* All preterm patients with a gestational age less than 37 weeks at the time of surgery.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nischal K Gautam, MD, Study Director — UTHealth
Locations (1):
- UT Health, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 enrolled participants declined to participate before being assigned to an intervention and therefore did not receive the intervention.
Period: Randomized Dosing (Doses 1 and 2)
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed
Started | 46 | 50
Received Dose 1 | 44 | 47
Received Dose 2 | 42 | 46
Completed | 42 | 46
Not Completed | 4 | 4
Not completed — Did not receive intervention because peripheral arterial line (PAL) was replaced due to spasm | 2 | 3
Not completed — Did not receive second dose | 2 | 1
Period: Rescue Papaverine (Optional Dose 3)
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed
Started (Only participants who had suboptimal waveforms after the first 2 randomized doses in the previous period went on to receive rescue papaverine in this period. 7 in the Papaverine plus Heparin arm received rescue papaverine. 17 in the Heparin arm received rescue papaverine.) | 7 | 17
Received Rescue Papaverine | 7 | 17
Completed | 7 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for all participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed | Total
Number analyzed (Participants) | 42 | 46 | 88
Age, Continuous [Mean (Standard Deviation); unit: months] | 24.1 (46.9) | 24.7 (39.5) | 24.5 (43.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 22 | 26 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 46 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Optimal Arterial Waveform
Description: Optimal waveform was defined as easy aspiration of a blood sample (negative aspiration is easy and draws back freely without cavitation, and takes no more than 30 seconds to draw 1 mL), absence of color change at the catheter insertion site, and presence of a dicrotic notch in the arterial pressure waveform (a distinct dicrotic notch implies system has good resolution at higher frequencies and is not overdamped).
Time Frame: 5 minutes after first dose
Population: These data were not collected for 2 participants in the Papaverine plus Heparin arm and 1 in the Heparin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed
Number analyzed (Participants) | 42 | 46
Participants | 27 | 18

2. Secondary Outcome: Number of Participants With Optimal Arterial Waveform
Description: as for outcome 1
Time Frame: 60 minutes after first dose
Population: These data were not collected for 2 participants in the Papaverine plus Heparin arm and 1 in the Heparin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed
Number analyzed (Participants) | 42 | 46
Participants | 30 | 28

3. Secondary Outcome: Number of Participants With Suboptimal Waveforms Who Received Rescue Papaverine and for Whom Papaverine Rescued Suboptimal Waveforms
Description: These data were collected only from participants who received rescue papaverine. 7 in the Papaverine plus Heparin arm received rescue papaverine. 17 in the Heparin arm received rescue papaverine.
Time Frame: 5 minutes after injection of rescue papaverine (about 70 minutes after first study drug dose and about 10 minutes after second study drug dose)
Population: These data were collected only from participants who received rescue papaverine. 7 in the Papaverine plus Heparin arm received rescue papaverine. 17 in the Heparin arm received rescue papaverine.
Measure: Count of Participants; unit: Participants
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed
Number analyzed (Participants) | 7 | 17
Participants | 3 | 13

ADVERSE EVENTS:
Time Frame: about 6 hours
Arm/Group | Papaverine Plus Heparin During Procedure, With Rescue Papaverine as Needed | Heparin During Procedure, With Rescue Papaverine as Needed
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/46
Other Adverse Events (participants affected / at risk) | 0/42 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03894904/Prot_001.pdf